CLINICAL TRIAL: NCT01867554
Title: Recherche et caractérisation de Nouveaux gènes impliqués Dans la déficience Intellectuelle.
Brief Title: Research and Characterization of New Genes Involved in Intellectual Disability
Acronym: GeneDefi
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C12-06; 2012-A00936-37 (Registry Identifier: IDRCB)
Record Dates: First submitted 2013-01-28; First posted 2013-06-04 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Intellectual Disability
Keywords: Intellectual disability; Autism spectrum disorders; gene; Next generation sequencing
MeSH Terms: conditions — Intellectual Disability; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA RNA Plasma Urines
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intellectual disability: patients with intellectual disability or psycho-motor retardation and their parents and sibs (affected or not)
  Interventions: Genetic: gene analysis

INTERVENTIONS:
Genetic: gene analysis — gene analysis

SUMMARY:
Intellectual disability (ID) occurs in 2 to 3 % of the general population but the cause is identified only in 30 to 60% of cases.

The purpose of this study is to indentify genes involved in ID with new genetics tools (SNP-arrays, next generation sequencing...) and establish genotype-phenotype correlations.

ELIGIBILITY:
Inclusion Criteria:

* for the patients: Clinical diagnosis of intellectual disbility
* for the unaffected sibs: to be aged at least 3 years
* informed consent

Exclusion Criteria:

* absence of informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * 2500 patients with intellectuel disability
  * 5000 parents or unaffected sibs
  * 1000 affected sibs
Sampling Method: Non-Probability Sample
Enrollment: 8500 (Actual)
Dates: Start 2012-12-31 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with genetic cause identified | 5 years
  Number of participants for which the causative gene of intellectual disability will be identified and number of genes involved in intellectual disability identified with new technologies including microarray and next generation sequencing

SECONDARY OUTCOMES:
genotype-phenotype correlations | genotype-phenotype correlations (according to the genes identified in a period of 5 years)
  Explore genotype-phenotype correlations when a new gene involved in intellectual disability will be identified

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Brice, MD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- CRICM - UPMC/Inserm UMR_S975/CNRS UMR7225, Groupe Hospitalier de la Pitié-Salpêtrière,, Paris, France

REFERENCES:
- [Background] Nava C, Lamari F, Heron D, Mignot C, Rastetter A, Keren B, Cohen D, Faudet A, Bouteiller D, Gilleron M, Jacquette A, Whalen S, Afenjar A, Perisse D, Laurent C, Dupuits C, Gautier C, Gerard M, Huguet G, Caillet S, Leheup B, Leboyer M, Gillberg C, Delorme R, Bourgeron T, Brice A, Depienne C. Analysis of the chromosome X exome in patients with autism spectrum disorders identified novel candidate genes, including TMLHE. Transl Psychiatry. 2012 Oct 23;2(10):e179. doi: 10.1038/tp.2012.102. PMID 23092983